CLINICAL TRIAL: NCT06286488
Title: Immunological and Clinical Effectiveness and Tolerability of Tetravalent Inactivated Influenza Vaccine in Patients at Risk for Severe and Complicated Influenza
Brief Title: Effectiveness and Tolerability of Influenza Vaccine in Patients at Risk for Severe and Complicated Influenza
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Principal Investigator, ANNA JAGIELSKA, Principal Investigator, Medical University of Warsaw
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KB/96/2020
Record Dates: First submitted 2024-02-22; First posted 2024-02-29 (Actual); Last update posted 2024-03-01 (Actual); Status verified 2024-02

CONDITIONS: Influenza; Obesity; Pregnancy; Infection; Elderly Infection; Vaccine Reaction; Vaccine Adverse Reaction; Tolerance
Keywords: influenza; vaccination; immunogenicity; efficacy; obesity; pregnancy
MeSH Terms: conditions — Influenza, Human; Obesity; Pregnancy Complications, Infectious | interventions — vaxigrip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Evaluation of immunogenicity and tolerance of quadrivalent influenza vaccine in obese adults (Experimental): Scientific observations published during the 2009 influenza pandemic have highlighted the more severe course and complications of influenza in obese people. The effect of excessive body fat in humans on the immune response to influenza vaccination is not fully explained by the available studies. Study aim was the evaluation of immunological efficacy and tolerance of QIV in obese adult patients and the relationship between the degree of obesity and immunogenicity of quadrivalent QIV in obese adult patients. Free of charge influenza vaccination was done with a quadrivalent Sanofi Pasteur Vaxigrip Tetra vaccine at a dose of 0.5 ml according to WHO recommendations for 2017/2018 for the northern hemisphere.
  Interventions: Drug: Vaxigrip
- Immunogenicity of QIV in pregnant women, including transplacental transport of antibodies (Experimental): Many studies confirm the safety of vaccinations against influenza during pregnancy for pregnant women as well for children. Previous studies have assessed the immunological efficacy of a monovalent and trivalent vaccine, but studies assessing the immunological efficacy and tolerability of the tetravalent, inactivated influenza vaccine in pregnant women are missing.The aim of the study is to assess immunogenicity and tolerance of tetravalent, inactivated influenza vaccine in pregnant women, depending on the duration of vaccination (II or III trimester) by assessing the level of antibodies in neonatal umbilical cord blood (transplacental transfer). Free of charge influenza vaccination was done with a quadrivalent Sanofi Pasteur Vaxigrip Tetra vaccine at a dose of 0.5 ml according to WHO recommendations for 2021/2022, 2022/2023 for the northern hemisphere.
  Interventions: Drug: Vaxigrip

INTERVENTIONS:
Drug: Vaxigrip — Evaluation of immunogenicity and tolerance of quadrivalent influenza vaccine in groups at risk of severe influenza, including obese adults, as well as in pregnant women (with assesment of antibodies in cord blood).

SUMMARY:
The aim of the study is to evaluate simultaneously the immunological and clinical efficacy and tolerability of an influenza vaccine, inactivated, quadrivalent, with cleaved virus, in patients at risk for severe and complicated influenza routinely vaccinated against influenza in family medicine clinics or specialty clinics (pediatric, internal medicine, cardiology, gynecological diabetes, pregnant women, transplant).

DETAILED DESCRIPTION:
Influenza has been called the last uncontrollable scourge of mankind because of its epidemic and pandemic potential. According to WHO estimates, 5-10% of the adult population and 10-20% of children globally fall ill with influenza seasonally. Influenza incidence has implications for individual patients (risk of complications, hospitalization, disability and death), as well as for public health (increased outpatient consultations, hospitalizations, including in intensive care units, increased absenteeism from work). Groups at risk for post-influenza complications include children under the age of 5, seniors over 65, patients with chronic diseases such as respiratory, cardiovascular, metabolic conditions, obesity, immunosuppressive treatment, and pregnant women, among others. Since the influenza A H1N1pdm09 pandemic, the WHO has particularly emphasized the need to vaccinate patients at risk of severe and complicated influenza, and has recommended a tetravalent vaccine since 2013. The inactivated tetravalent influenza vaccine has been available in Poland since the 2016/17 season, and also registered for children since the 2018/19 season. This is also in line with current Polish recommendations issued by the National Influenza Control Program. With the extremely low level of vaccination against influenza of the Polish population (about 3.7%), the threat of an influenza epidemic is serious. The number of reports describing simultaneously the immunological and clinical efficacy and tolerance of influenza vaccination of the Polish population is limited, the published works usually focus on the evaluation of either immunogenicity or clinical efficacy, there is a lack of publications comprehensively determining the effectiveness of the vaccine in the Polish homogeneous population, especially people in the above-mentioned risk groups, as well as the determination of the occurrence of the phenomenon of non-immunogenicity of the vaccine in the Polish population. An important aspect in the situation of low immunogenicity of the Polish population is the aspect of persistence of protective antibody levels at the beginning of the next flu season. Few works indicate the persistence of protective antibody levels in healthy individuals without risk factors for immune disorders, but the quality of "immune memory" after influenza vaccination in patients at risk of severe and complicated influenza is still insufficiently understood.

The aim of the study is to evaluate simultaneously the immunological and clinical efficacy and tolerability of an influenza vaccine, inactivated, quadrivalent, with cleaved virus, in patients at risk for severe and complicated influenza routinely vaccinated against influenza in family medicine clinics or specialty clinics (pediatric, internal medicine, cardiology, gynecological diabetes, pregnant women, transplant).

ELIGIBILITY:
Inclusion criteria for the study:

1. age over 18 (adults able to give informed consent to participate in the study) or age under 18 and the consent of a legal guardian and, in the case of persons aged 16-18, also the consent of a minor;
2. belonging to groups at risk of severe and complicated course of influenza (children, elderly people, patients with chronic diseases, pregnant women);
3. no clinical contraindications to influenza vaccination;
4. the patient and/or his legal guardians give written, informed consent to participate in the study.

Exclusion criteria from the study:

1. lack of consent to participate in the study - at every stage of the study;
2. clinical contraindications to influenza vaccination.

Clinical contraindications to influenza vaccination:

* exacerbation of a chronic disease;
* acute infectious disease;
* allergy to a vaccine component;
* a serious allergic reaction after a previous flu vaccination;
* Guillain-Barre syndrome up to 6 weeks after the previous vaccination;
* use of immunosuppressive treatment (relative contraindication)

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — In the arm concerning pregnant patients, only women
Enrollment: 1500 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
influenza vaccine immunogenicity, seroconversion and seroprotection | 4-8 weeks after vaccination
  Immunogenicity is assessed using a hemagglutinin inhibition test. Percentage of patients with influenza antibody titers of 1:40 or more after vaccination. Seroconversion rate-a fourfold increase in the geometric mean titer after vaccination and the percentage of newborns with antibody titers of 1:40 or more at birth. Seroconversion and seroprotection were compared against the second and third trimesters of pregnancy. Transplacental transfer of antibodies was compared according to whether or not the patient had been vaccinated in previous seasons (applies only to the study on pregnant women.

SECONDARY OUTCOMES:
assessment of vaccination tolerance | 30 days after vaccination
  Each patient will keep a diary of symptoms of adverse events occurring after vaccination and after 4 weeks will be asked to complete a survey (the survey was created in accordance with the Summary of Product Characteristics, CPMP and International Committee for Harmonization guidelines for the management of clinical safety data: definitions and standards for accelerated reporting).

CONTACTS AND LOCATIONS:
Overall Officials: Monika Zasztowt-Sternicka, MD, Principal Investigator — Doctoral School, Medical University of Warsaw
Locations (1):
- Department of Social Medicine and Public Health, Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zasztowt-Sternicka M, Jagielska A, Rzad M, Szymusik I, Hallmann E, Brydak L, Nitsch-Osuch A. Immunogenicity of inactivated quadrivalent influenza vaccine in pregnant women, including the level of postvaccination antibodies in umbilical cord blood. Vaccine. 2025 Apr 19;53:127047. doi: 10.1016/j.vaccine.2025.127047. Epub 2025 Apr 8. PMID 40203592